CLINICAL TRIAL: NCT04844814
Title: Anakinra vs Prednisone to Treat Gout Flare in Patients With Chronic Kidney Disease Stage 4/5 or Renal Transplantation: a Randomized, Double Blinded, Multicenter Study
Brief Title: Anakinra vs Prednisone to Treat Gout Flare in Patients With Chronic Kidney Disease Stage 4/5 or Renal Transplantation
Acronym: Ana4CKD
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Peremption of treatments, difficulty of patients recrutment (28 patients in 3 years) and lack of funding to pursue the study.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP180560
Record Dates: First submitted 2021-01-24; First posted 2021-04-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Gout; Chronic Kidney Disease; Renal Transplantation
Keywords: Gout; Flare; Urate crystals; Chronic kidney disease; Anakinra; IL-1b; Corticosteroid; Renal transplantation
MeSH Terms: conditions — Gout; Renal Insufficiency, Chronic | interventions — Interleukin 1 Receptor Antagonist Protein; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anakinra (Experimental): Anakinra 100 mg/d+Placebo of Prednisone
  Interventions: Drug: Anakinra 100Mg/0.67Ml Inj Syringe; Drug: Placebo of Prednisone
- Prednisone (Active Comparator): Prednisone 30 mg/d+Placebo of Anakinra
  Interventions: Drug: Prednisone; Drug: Placebo of Anakinra

INTERVENTIONS:
Drug: Anakinra 100Mg/0.67Ml Inj Syringe — Anakinra 100 mg/d subcutaneous injection
  Arms: Anakinra
Drug: Prednisone — Prednisone 30 mg/d
  Arms: Prednisone
Drug: Placebo of Prednisone — Placebo of Prednisone
  Arms: Anakinra
Drug: Placebo of Anakinra — Placebo of Anakinra
  Arms: Prednisone

SUMMARY:
Gout is secondary to urate crystal deposition after chronic elevation of serum urate level. Urate crystal deposition is responsible for acute and recurrent inflammatory flares which can be treated with colchicine, non-steroid anti-inflammatory drugs (NSAID), corticosteroid or interleukin (IL)-1b blockade. Colchicine and NSAID are contra-indicated in patients with chronic renal disease (CKD) stage 4/5 or with renal transplantation. In these patients gout flare is treated with high dose of corticosteroid or IL-1b inhibitors.

Frequent use of high dose of corticosteroid can worsen gout comorbidities including mellitus diabetes type 2, hypertension, obesity and dyslipidemia. Anakinra, an IL-1b receptor antagonist, is efficient in gout flare in patients without CKD stage 4/5.

The aim of this study is to demonstrate that anakinra is superior to prednisone to treat gout flare in patients with CKD 4/5 or renal transplantation.

DETAILED DESCRIPTION:
The study will include 234 gouty patients with CKD 4/5 or renal transplantation with gout flare

This study will include the following visits:

- Selection/inclusion visit (V0):

Patient with gout flare and CKD 4/5 or renal transplantation will be included and randomized to receive either anakinra 100 mg/d or prednisone 30 mg/d.

-Visit from day (d)0 to d5: included patients will be hospitalized and treatment will be administrated by a nurse. Treatment will be stopped if patient had ≥ 80% improvement. Treatment response is defined by improvement ≥ 50%.

Patient will be evaluated every day from d0 to d5. At d3, if improvement is < 50%, patient will be considered as non-responder and patient will be managed as physician's habits.

At d5, if improvement is < 80%, patient will be managed as physician's habits Between d1 and d5, if improvement ≥ 80%, patient can be discharged and will have a visit at d5 as outpatient.

- Visit month (M)1 end of research: clinical evaluation of gout, demographic characteristics, medication, number of gout flare within the month, number of hospitalization and/or medical consultation within the month, blood analysis (serum creatinine level, eGFR, SUL, CRP, HbA1C, total, HDL and LDL cholesterol, triglyceride, glycaemia).

The study ends after the M1 consultation. The total duration of participation in the study is 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18 years old
* Gout confirmed by identification of urate crystals by joint fluid or tophus analysis or by ultrasound of the affected joint and/or
* Gout according to Nijmegen criteria (presence of a score ≥ 8/13) depending on the following items:

Man (2 pts) Previous crisis (2 pts) Involvement of first metatarsophalangeal joint (MTP1) (2.5 pts) Maximum pain within 24 hours (0.5pt) Redness (1 pt) HTA or cardiovascular disease (1.5 pts) SUL > 360 μmol/l during the crisis (3.5 pts)

* Chronic kidney disease stage 3b/4/5 or renal transplantation
* Flare ≤ 5 days
* Pain assessed by visual analogical scale > 4/10

Exclusion Criteria:

* Participating in another trial including the administration of a drug
* Active infection
* History of anakinra or prednisone allergy
* Contra-indication of anakinra or prednisone
* Neutrophil count < 1000/mm3 (not due to ethnic cause)
* Difficulty understanding French
* Illiteracy
* Pregnant women or breastfeeding mothers (see PHC article L.1121-5)
* Persons deprived of liberty by judicial or administrative decision, persons receiving psychiatric care under Sections L. 3212-1 and L. 3213-1 and persons admitted to a health or social institution for purposes other than research (see CSP Article L.1121-6)
* Major persons subject to a measure of legal protection or unseeding to express consent (see PHC Article L.1121-8)
* Persons not affiliated to a social security plan or beneficiaries of such a plan (see PHC Article L.1121-8-1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain difference between Day 3 and treatment initiation | Day 3
  Pain difference between day 3 and treatment initiation assessed by visual analogical scale (VAS) from 0 to 10 VAS = 0, no pain VAS =10, maximal pain

SECONDARY OUTCOMES:
Percentage of responders (improvement ≥ 50%) at day 5 | Day 5
  Percentage of responders (improvement ≥ 50%) at day 5
Percentage of flare resolution (improvement ≥ 80%) at day 5 | Day 5
  Percentage of flare resolution (improvement ≥ 80%) at day 5
Time to treatment response | Day 3 or Day 5
  Time to treatment response
Time to flare resolution | Day 3 or Day 5
  Time to flare resolution
Treatment duration | Day3 or Day 5
  Treatment duration
Duration of hospitalization | Day 3 or Day 5
  Duration of hospitalization
Healthcare consumption at month 1 : number of consultations and hospitalizations related to gout flare | Month 1
  Healthcare consumption at month 1 assessed by number of consultations and hospitalizations related to gout flare
Healthcare consumption at month 1: total hospital stay | Month 1
  Healthcare consumption at month 1 assessed by total hospital stay
Healthcare consumption at month 1 | Month 1
  Healthcare consumption at month 1 assessed by number and cumulative duration of sick leave related to gout
Side effects | Month 1
  Side effects
Comorbidity decompensations at month 1 : DT2 decompensation | Month 1
  Comorbidity decompensations at month 1 assessed by DT2 decompensation measure
Comorbidity decompensations at month 1: Blood pressure | Month 1
  Comorbidity decompensations at month 1 assessed by Blood pressure measure
Comorbidity decompensations at month 1: Hypertension | Month 1
  Comorbidity decompensations at month 1 assessed by hypertension measure
Comorbidity decompensations at month 1: Weight | Month 1
  Comorbidity decompensations at month 1 assessed by Weight measure
Comorbidity decompensations at month 1: number of Cardiovascular events : coronary disease, heart attack, stroke | Month 1
  Comorbidity decompensations at month 1 assessed by number of Cardiovascular events : coronary disease, heart attack, stroke
Comorbidity decompensations at month 1: Blood analysis of serum creatinine level | Month 1
  Comorbidity decompensations at month 1 assessed by serum creatinine level measure
Comorbidity decompensations at month 1: Blood analysis of epidermal Growth Factor Receptor (eGFR) | Month 1
  Comorbidity decompensations at month 1 assessed by eGFR measure
Comorbidity decompensations at month 1: Blood analysis of C reactive protein (CRP) | Month 1
  Comorbidity decompensations at month 1 assessed by CRP measure
Comorbidity decompensations at month 1: Blood analysis of HbA1C | Month 1
  Comorbidity decompensations at month 1 assessed by HbA1C measure
Comorbidity decompensations at month 1: Blood analysis of total cholesterol | Month 1
  Comorbidity decompensations at month 1 assessed by total cholesterol measure
Comorbidity decompensations at month 1: Blood analysis of LDL cholesterol | Month 1
  Comorbidity decompensations at month 1 assessed by HDL cholesterol measure
Comorbidity decompensations at month 1: Blood analysis of HDL cholesterol | Month 1
  Comorbidity decompensations at month 1 assessed by HDL cholesterol measure
Comorbidity decompensations at month 1: Blood analysis of triglyceride | Month 1
  Comorbidity decompensations at month 1 assessed by triglyceride measure
Comorbidity decompensations at month 1: Blood analysis of glycaemia | Month 1
  Comorbidity decompensations at month 1 assessed by glycaemia measure
site injection reaction during day 0 to day 5: pain | Dat 3 or day 5
  site injection reaction during day 0 to day 5 assessed by pain (0-10 scale VAS) measure
site injection reaction during day 0 to day 5: inflammatory reaction | Dat 3 or day 5
  site injection reaction during day 0 to day 5 assessed by CRP level measure
site injection reaction during day 0 to day 5: swelling (yes/no) | Dat 3 or day 5
  site injection reaction during day 0 to day 5 assessed by swelling (yes/no)
site injection reaction during day 0 to day 5: itching (yes/no) | Dat 3 or day 5
  site injection reaction during day 0 to day 5 assessed by itching (yes/no)
site injection reaction during day 0 to day 5: redness (yes/no) | Dat 3 or day 5
  site injection reaction during day 0 to day 5 assessed by redness (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Hang-Korng EA, PhD-MD, Principal Investigator — Hôpital Lariboisière
Locations (1):
- Rhumathology department, Paris, Île-de-France Region, France